CLINICAL TRIAL: NCT03717571
Title: ROTCUFF - Measuring Load-induced Superior Glenohumeral Translation in Patients With Degenerative Rotator Cuff Tears and Asymptomatic Subjects: 3-dimensional Motion Analysis Versus Single Plane Fluoroscopy
Brief Title: Superior Glenohumeral Translation in Patients With Degenerative Rotator Cuff Tears
Acronym: ROTCUFF
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2018-01692
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: age and sex matched healthy control persons
  Interventions: Diagnostic Test: Glenohumeral translation assessment
- isolated tear: patients with isolated complete supraspinatus muscle tear
  Interventions: Diagnostic Test: Glenohumeral translation assessment
- combined tear: patients with complete supraspinatus muscle tear and either partial infraspinatus muscle tear or partial subscapularis muscle tear
  Interventions: Diagnostic Test: Glenohumeral translation assessment

INTERVENTIONS:
Diagnostic Test: Glenohumeral translation assessment — amount of glenohumeral translation under load

SUMMARY:
Degenerative partial and complete rupture of the rotator cuff is a common injury among elder patients. However, the clinical manifestation varies largely with some patients having severe pain and limiting range of motion and others having no complaints. The basic functions of the rotator cuff are to facilitate shoulder motion and stabilization and centering of the glenohumeral joint. The objective of this study is to quantify the difference in superior glenohumeral translation in patients with degenerative rotator cuff tear compared to healthy control subjects and to determine the effect of isolated complete supraspinatus tear and combined complete supraspinatus and either partial infraspinatus or partial subscapularis tear.

DETAILED DESCRIPTION:
The study will examine a cohort of 10 patients with isolated complete supraspinatus muscle tear and 10 patients with complete supraspinatus muscle tear and either partial infraspinatus muscle tear or partial subscapularis muscle tear, and a cohort of 10 age-matched healthy control persons. The participants will be recruited from the Clinic of Orthopaedics and Traumatology at the University Hospital Basel. Inclusion criteria: 45 years < age < 65 years; degenerative complete supraspinatus muscle tear or complete supraspinatus muscle tear and either partial infraspinatus muscle tear or partial subscapularis muscle tear; unilateral rotator cuff tear. Exclusion criteria: traumatic tendon ruptures; prior treatment of the ipsilateral upper extremity; clinical history of the contralateral glenohumeral joint; no complete supraspinatus muscle tear; tears in more than two rotator cuff muscles; neuromuscular disorders affecting upper limb movement; additional pathologies that influence the mobility of the shoulder joint; inability to provide informed consent.

Patients will complete the health questionnaire and reflective markers and electromyographic sensors will be placed on anatomical landmarks and shoulder muscles, respectively, before loaded and unloaded abduction and flexion arm movements will be performed. Centre of rotation of both shoulders will be calculated to determine glenohumeral translation. This parameter will be compared between patient groups and control subjects using linear mixed models with group membership and load as fixed factor and subject as random factor. The critical shoulder angle will be included as covariate into the model to detect a potential modulating role of this factor on glenohumeral translation.

ELIGIBILITY:
Inclusion criteria patients

* 45 years ≤ age ≤ 65 years
* Degenerative complete supraspinatus muscle tear or complete supraspinatus muscle tear and either partial infraspinatus muscle tear or partial subscapularis muscle tear
* Unilateral rotator cuff tear

Exclusion criteria patients

* Traumatic tendon ruptures
* Incomplete supraspinatus muscle tear
* Tears in more than two rotator cuff muscles
* Prior conservative treatment or surgery of the ipsilateral upper extremity
* Clinical history of the contralateral glenohumeral joint
* Range of motion < 90° in abduction and flexion
* Neuromuscular disorders affecting upper limb movement
* Additional pathologies that influence the mobility of the shoulder joints
* Inability to provide informed consent

Inclusion criteria healthy control subjects

• 45 years ≤ age ≤ 65 years

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 10 patients with isolated complete supraspinatus muscle tear
  * 10 patients with complete supraspinatus muscle tear and either partial infraspinatus muscle tear or partial subscapularis muscle tear
  * 10 healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Glenohumeral translation | Baseline
  Amount of glenohumeral translation under load

SECONDARY OUTCOMES:
Disabilities of arm, shoulder and Hand (DASH) | Baseline
  assessed using the Quick DASH (0 - no problems, 100 - extreme problems)
Shoulder function | Baseline
  assessed using the Constant Shoulder Score (0 - no problems, >30 extreme problems)
Shoulder pain | Baseline
  assessed using a 15 cm visual analogue scale converted to 0 to 100 scale (0 - no pain; 100 - worst pain imaginable)
Critical shoulder angle (CSA) | Baseline
  measured on frontal plane radiographs in neutral arm position available from the clinical consultation. The CSA is the angle between the line connecting the superior with the inferior border of the glenoid fossa and the line connecting the inferior border of the glenoid fossa with the most inferolateral point of the acromion
Muscle activity | Baseline
  root mean square of the electromyography (EMG) signal during the arm movements calculated and normalised to the maximal obtained signal intensity
Glenohumeral translation from fluoroscopy | Baseline
  the perpendicular distance of the centre of the glenohumeral joint and the x-axis of the scapula coordinate system will be measured. Glenohumeral translation will be defined as the difference in this distance between the abducted arm positions and the resting arm position

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided